CLINICAL TRIAL: NCT07161323
Title: Comparison of the Acute Effects of Sustained Natural Apophyseal Glide and Sciatic Nerve Mobilization Exercises in Non-Specific Sciatic Nerve Pain
Brief Title: SNAG and SNME in Non-Specific Sciatic Pain
Acronym: CASE-SNAG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Çiçek Günday, Asst. Prof., Istinye University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 28032025
Record Dates: First submitted 2025-07-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Sciatica Pain; Sciatica Acute; Mulligan Mobilization
Keywords: Sciatic Nerve Pain; Mulligan Concept; Manual Therapy; Pain Management; Non-Specific Sciatica
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan Consept Group (MCG) (Experimental)
  Interventions: Other: Sustained Natural Apophyseal Glide (SNAG)
- Neural Mobilization Group (NMG) (Experimental)
  Interventions: Other: Sciatic Nerve Mobilization Exercises (SNME)

INTERVENTIONS:
Other: Sustained Natural Apophyseal Glide (SNAG) — In this intervention, participants will initially receive the SNAG technique targeting the L5-S1 lumbar segment. Participants will be seated on a treatment table with feet flat and knees at 90°. The therapist will position a specialized Mulligan belt around the L5-S1 segment and anchor it around their pelvis to generate a gentle traction force via controlled hip movement. While this force is applied, participants will perform active trunk flexion, holding the end-range position for 30 seconds. This movement will be repeated six times, constituting a 3-minute set. A total of 4 sets will be administered, with 2-minute rest periods between sets.
  Arms: Mulligan Consept Group (MCG)
Other: Sciatic Nerve Mobilization Exercises (SNME) — Participants will sit with hips and knees at 90° flexion, feet flat on the floor. The involved leg will be fully extended at the knee. In this position, the participant will be asked to perform ankle dorsiflexion and neck extension simultaneously (applying tension to the distal part of the sciatic nerve while relaxing the proximal part) and hold for 3 seconds. Next, the participant will plantarflex the ankle and flex the neck (tensioning the proximal end while relaxing the distal), again holding for 3 seconds. This 6-second sequence will be repeated 10 times per set. The exercise will be performed in 3 sets per leg, with 3-minute rests between sets.
  Arms: Neural Mobilization Group (NMG)

SUMMARY:
This study is designed as a crossover trial. All participants who meet the inclusion criteria and voluntarily agree to participate will be evaluated using the assessment methods detailed below. Subsequently, participants will be randomly assigned into two groups. The first group (Mulligan Concept Group - MCG) will receive the SNAG technique, while the second group (Neural Mobilization Group - NMG) will perform the Sciatic Nerve Mobilization Exercise (SNME). After the intervention, participants will be evaluated a second time. Ten days after this session, participants will be invited back. Those who were in the MCG group during the first session will be re-evaluated and then receive the SNGE intervention. Participants who were in the SNGE group during the first session will be re-evaluated and then receive the SNAG intervention. Following this second intervention, participants will be evaluated once again.

Assessments will be done are Demographic Form, Visual Analogue Scale, Oswestry Disability Index, Joint Range of Motion, Five-times Sit-to-stand Test, Sit and Reach Test

DETAILED DESCRIPTION:
The sciatic nerve, formed by the union of five spinal nerve roots (L4, L5, S1, S2, and S3), is one of the largest and most important peripheral nerves, carrying both motor and sensory fibers. Due to its complex anatomical course and position, sciatic nerve pain is a common form of neuropathic pain. Despite its high prevalence, research on the effectiveness of non-pharmacological treatments remains limited, restricting the development of evidence-based clinical guidelines for primary care management. One such conservative approach is sciatic nerve mobilization, also known as neurodynamic techniques or nerve gliding exercises. Sciatic Nerve Mobilization Exercises (SNME) aim to facilitate gentle sliding of the sciatic nerve along its anatomical pathway without overstretching or irritating it, thereby reducing pain and improving function. On the other hand, the Mulligan Concept (MC) is a modern manual therapy approach incorporating sustained natural apophyseal glides (SNAGs), especially effective for spinal dysfunctions. These mobilizations are typically pain-free and performed in conjunction with active patient movement. SNAGs target the lumbar spine to restore joint mechanics and relieve pain. Widely adopted in clinical practice, this method is used by a significant number of physiotherapists in the UK and US, often as part of their routine patient care. While both SNME and SNAGs are commonly used for managing non-specific sciatic pain, direct comparisons of their clinical efficacy are scarce. Therefore, this study aims to fill that gap by evaluating and comparing the acute effects of these two interventions in individuals with non-specific sciatic nerve pain. The objectives are to determine which technique is more effective in reducing pain, enhancing functional mobility, and improving daily activity performance. The study also seeks to assess which intervention yields better outcomes in terms of range of motion, functional movement, and flexibility. The null hypothesis (H0) posits no significant difference between SNME and SNAGs in improving pain and function in patients with non-specific sciatic pain, whereas the alternative hypothesis (H1) suggests a significant difference between the two. This research holds clinical relevance in guiding physiotherapists toward evidence-based interventions tailored to the needs of individuals suffering from this widespread and disabling condition.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 20 and 50,
* Individuals describing non-specific sciatic pain characterized by unilateral low back pain accompanied by radiating symptoms to the leg,
* Duration of pain longer than 12 weeks,
* Presence of pain during the Slump Test and Straight Leg Raise Test,
* No history of any physical therapy or intervention in the past month.

  b: Exclusion Criteria:
* Individuals diagnosed with herniated disc or spinal stenosis by a physician,
* Physician-diagnosed secondary neurological conditions,
* History of spinal surgery,
* Individuals describing the origin of their pain as the lower back (without leg involvement),
* Presence of neurological symptoms (e.g., foot drop, significant muscle weakness),
* Serious medical conditions that may affect treatment or outcomes (e.g., cancer, infections, or inflammatory diseases),
* Pregnancy or recent childbirth (within the past year),
* Use of medications that may affect pain perception or mobility (e.g., opioids),
* Inability to comply with the weekly treatment schedule.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | Through study completion, an average of 1 year
  The ODI assesses the impact of sciatic nerve pain on daily activities, including sitting, standing, walking, sleeping, and personal care. The total score indicates the level of disability.
5 Times Sit to Stand Test | Through study completion, an average of 1 year
  The test will be used to measure the time it takes for an individual to rise from a seated position and sit back down. The participant is prepared in a seated position on a standard chair with a height of 43-46 cm, with their back against the chair and arms crossed over the chest. Upon the command to begin, the participant stands up fully and then completes the test by sitting down and standing up a total of five times as quickly as possible.
Sit and Reach Test | Through study completion, an average of 1 year
  The participant will sit on a mat placed on a flat surface, with legs extended straight forward and knees fully extended. The soles of the feet will be positioned vertically and kept stable. The participant will then reach forward with both arms, aiming to touch the toes or reach beyond them if possible. The reach distance will be recorded in centimeters based on how far the fingertips are from the soles of the feet.

SECONDARY OUTCOMES:
Range of Motion | Through study completion, an average of 1 year
  Spinal flexion, extension, and lateral flexion range of motion (ROM) will be assessed using a goniometer. The patient will be prepared in an upright standing position, with feet shoulder-width apart, arms relaxed at the sides, and maintaining a straight posture. Then the function will be done by the patient actively.
Pain Intensity Visual Analog Scale (VAS) | Through study completion, an average of 1 year
  Pain intensity will be evaluated using the Visual Analog Scale (VAS), where participants rate their pain from 0 (no pain) to 10 (worst imaginable pain). Pain will be measured during sitting, forward bending, and walking, for both back and leg pain.

CONTACTS AND LOCATIONS:
Overall Officials: Çiçek Günday, Asst.Prof., Principal Investigator — Istinye University; Sohiab Hassan Mohamed Wagdy Ahmed Elsayed Eladawi, Physiotherapist, Study Chair — Istinye University
Locations (1):
- Clam Fizyoterapi Merkezi, Istanbul, Turkey (Türkiye)